CLINICAL TRIAL: NCT06735131
Title: A Prospective, Multicenter Clinical Trial Exploring the Optimal Combination Strategies of Radiotherapy and Immunotherapy for Advanced Triple-Negative Breast Cancer
Brief Title: The Optimal Radioimmunotherapy Combinations for Advanced TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: West China Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-025
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Triple-Negative Breast Cancer (TNBC)
Keywords: radiotherapy; immunotherapy; chemotherapy; triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1: 5Gy × 5 , daily (Experimental): within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Interventions: Radiation: radiotherapy 5 Gy × 5 fractions, once a day; Drug: Toripalimab; Drug: chemotherapy regimen selected by the investigator
- Arm 2: 8Gy × 5 , daily (Experimental): within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Interventions: Radiation: radiotherapy 8 Gy × 5 fractions, once a day; Drug: Toripalimab; Drug: chemotherapy regimen selected by the investigator
- Arm 3: 8Gy × 3, every other day (Experimental): within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Interventions: Radiation: radiotherapy 8 Gy × 3 fractions, once every other day; Drug: Toripalimab; Drug: chemotherapy regimen selected by the investigator
- Arm 4: 10Gy × 3, every other day (Experimental): within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Interventions: Radiation: radiotherapy 10 Gy× 3 fractions, once every other day; Drug: Toripalimab; Drug: chemotherapy regimen selected by the investigator
- Arm 5: 0.5Gy twice-a-day × 2 days, repeat for 4 cycles (8 Gy in total) (Experimental): on the first 2 days of first 4 cycles of toripalimab and chemotherapy
  Interventions: Radiation: radiotehrapy 0.5Gy twice-a-day × 2 days, repeat for 4 cycles (total 8Gy); Drug: Toripalimab; Drug: chemotherapy regimen selected by the investigator

INTERVENTIONS:
Radiation: radiotherapy 5 Gy × 5 fractions, once a day — 5 Gy × 5 fractions, once a day, beginning on the day within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Arms: Arm 1: 5Gy × 5 , daily
Radiation: radiotherapy 8 Gy × 5 fractions, once a day — 8 Gy × 5 fractions, once a day, beginning on the day within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Arms: Arm 2: 8Gy × 5 , daily
Radiation: radiotherapy 8 Gy × 3 fractions, once every other day — 8 Gy × 3 fractions, once every other day, beginning on the day within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Arms: Arm 3: 8Gy × 3, every other day
Radiation: radiotherapy 10 Gy× 3 fractions, once every other day — 10 Gy × 3 fractions, once every other day, beginning on the day within 4 weeks before the initiation of cycle of toripalimab and chemotherapy
  Arms: Arm 4: 10Gy × 3, every other day
Radiation: radiotehrapy 0.5Gy twice-a-day × 2 days, repeat for 4 cycles (total 8Gy) — 0.5 Gy twice-a-day × 2 days, on the first 2 days of the first 4 cycles of toripalimab and chemotherapy (total 8Gy)
  Arms: Arm 5: 0.5Gy twice-a-day × 2 days, repeat for 4 cycles (8 Gy in total)
Drug: Toripalimab — Toripalimab (240 mg IV, d1, Q3W)
Drug: chemotherapy regimen selected by the investigator — Regimens to be selected from: (1) Nab-paclitaxel (125 mg/m2 IV, days 1, 8, Q3W) (2) Gemcitabine (1000 mg/m² IV, days 1 and 8, Q3W) + carboplatin (AUC=2 IV, days 1 and 8, Q3W)

SUMMARY:
This study aims to explore the best combination patterns of radiotherapy and immunotherapy for advanced triple-negative breast cancer (TNBC).

DETAILED DESCRIPTION:
Metastatic triple-negative breast cancer (mTNBC) is a particularly aggressive form of breast cancer that poses significant therapeutic challenges. Because mTNBC tumors do not express estrogen receptors (ER), progesterone receptors (PR), or HER2, patients with this subtype cannot receive benefits from endocrine therapy or HER2-targeted treatments, leaving chemotherapy as the main treatment option. However, the effectiveness of traditional chemotherapy drugs is limited and they often come with severe side effects. This leads to short durations of progression-free survival (PFS) and overall survival (OS), and the development of drug resistance, which can cause the cancer to recur and spread.

Recently, the advent of immune checkpoint inhibitors has offered new therapeutic prospects for mTNBC. Inhibitors of PD-1/PD-L1, such as Pembrolizumab, Atezolizumab, and Toripalimab, have demonstrated some effectiveness in clinical trials, especially in patients with PD-L1-positive tumors. Yet, the overall response to immunotherapy remains low, and there is a risk of immune-related adverse events (irAEs), which require vigilant monitoring.

To address the shortcomings of both chemotherapy and immunotherapy, researchers are investigating innovative treatment strategies. These include targeting additional immune checkpoint molecules within the tumor microenvironment, developing novel chemotherapy drugs, and integrating immunotherapy with other treatments like radiotherapy. Local radiotherapy can substantially stimulate the immune system, increasing the antigenicity of cancer cells and enhancing the ability of cytotoxic T lymphocytes to recognize and attack cancer cells.

Although combined radiotherapy and immunotherapy have shown promise in treating other types of cancer, the most effective combination patterns, optimal radiotherapy dosing schedules, and the most suitable patient groups for advanced breast cancer, particularly mTNBC, are not well defined. This study seeks to identify the best combinations of radiotherapy and immunotherapy for advanced breast cancer, with the aim of improving survival rates and setting new standards for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable locally advanced/metastatic triple-negative breast cancer (defined as ER and PR <1%; and HER2 negative as IHC 0 or IHC 1+, or IHC 2+ but negative upon fluorescence in situ hybridization (FISH) testing). Patients with ER/PR ≤10% and deemed unsuitable for endocrine therapy by the investigator are also eligible.
2. No prior chemotherapy for advanced/metastatic disease.
3. ECOG PS score of 0 or 1.
4. Presence of 1 to 5 tumor lesions suitable for radiotherapy (individual lesion size between 0.5 and 5 cm, not limited to 1 to 2 organs).
5. At least one measurable lesion outside the radiation field that can be evaluated.
6. Suitable to receive one of the chemotherapy regimens chosen by the investigator: nab-paclitaxel or gemcitabine + carboplatin.
7. Patients with brain metastases are allowed if they do not require local therapy at enrollment or if the metastatic lesion is treated with the assigned radiotherapy regimen.
8. Patients who have previously received PD-1/PD-L1 therapy for early-stage disease are allowed to enroll.
9. Able to provide tumor tissue sections or agree to tumor biopsy during the screening period.
10. Adequate organ and bone marrow function, with specific requirements:

    1. Hematology: Neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥90×10^9/L; Hemoglobin (Hb) ≥90 g/L; No blood product transfusion (including red blood cell and platelet products, etc.) or growth factor (including colony-stimulating factors, interleukins, and erythropoietin, etc.) support treatment within 2 weeks prior to examination.
    2. Liver function: Serum total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5×ULN (for patients with liver metastases: ALT and AST ≤5×ULN).
    3. Renal function: Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance >60 mL/min.

Exclusion Criteria:

1. Received platinum-containing regimens during the adjuvant/neoadjuvant therapy phase, and the interval from the last treatment to recurrence/metastasis is less than 6 months.
2. Have received radiotherapy within 12 weeks prior to enrollment, unless the radiotherapy was for adjuvant purposes and there are lesions outside the previously irradiated field.
3. Extensive tumor metastasis with surrounding normal tissues that cannot tolerate radiotherapy damage.
4. Significant third-space fluid retention (e.g., ascites, pleural effusion, pericardial effusion).
5. Require long-term systemic corticosteroid treatment.
6. Have active autoimmune diseases.
7. Have concurrent severe infections.
8. Other patients deemed unsuitable for enrollment by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 6 months (6m-PFS rate) | 6 months
  Progression-free survival at 6 months (6m-PFS rate) is defined as the percentage of patients who have not experienced disease progression or death due to any cause at the 6-month mark after starting treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  Progression-free survival (PFS) is defined as the time from treatment initiation to disease progression or death from any cause.
Overall survival (OS) | up to 3 years
  Overall survival (OS) is defined as the time from treatment initiation to death from any cause.
Objective Response Rate | up to 3 years
  Objective response rate (ORR) is defined as the percetage of patients achieving a complete response (CR) or partial response (PR) according to RECIST v.1.1.
Duration of response | up to 3 years
  Duration of response (DOR) is defined as the duration from response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first.
Number of participants with treatment-related adverse events | up to 3 years
  Adverse events are assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No